CLINICAL TRIAL: NCT00525213
Title: A Phase II, Randomised, Double-blind, International, Multicentre, Placebo-controlled, Dose-ranging, Parallel-group Study to Evaluate the Efficacy and Safety of Orally Administered Rob 803 When Added to Stable Methotrexate
Brief Title: Study to Evaluate the Efficacy and Safety of Orally Administered Rob 803 When Added to Methotrexate
Acronym: ROBUST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: OxyPharma (Industry)
Responsible Party: Ulf Björklund, OxyPharma AB
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2006-004834-33
Record Dates: First submitted 2007-09-04; First posted 2007-09-05 (Estimated); Last update posted 2009-08-21 (Estimated); Status verified 2009-08

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — 9-chloro-2,3-dimethyl-6-(N,N-dimetylamino-2-oxoethyl)-6H-indolo(2,3-b)quinoxaline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- A (Active Comparator)
  Interventions: Drug: Rob 803
- B (Active Comparator)
  Interventions: Drug: Rob 803
- C (Active Comparator)
  Interventions: Drug: Rob 803
- D (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rob 803 — two capsules per day during 12 weeks
  Arms: A; B; C
Drug: Placebo — two capsules per day during 12 weeks
  Arms: D

SUMMARY:
The primary objective of this study is to evaluate the efficacy (ACR20) of Rob 803 administered orally once daily for 12 weeks in combination with a stable dose of methotrexate in subjects with moderate or severe active RA.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a common, chronic, disabling systemic autoimmune disease in which inflammation of the joint lining (synovium) occurs when the body's tissues are attacked by the immune system. The joint inflammation begins in the synovium and slowly destroys the cartilage, narrowing the joint and eventually damaging the bone. A large amount of inflammatory mediators or rheumatoid factors are synthesised in the joint which accelerate proliferation and differentiation of immune cells further to amplify the autoimmune reaction. A widely accepted model has emerged in which the presence of inflammation in established RA is driven by interactions between T cells, macrophages, and fibroblasts in an abnormal microenvironment.

Rheumatoid arthritis has an annual incidence of approximately 0.2 per 1000 in males and 0.4 per 1000 in females. In general, higher rates have been reported in the USA than in European populations. The incidence of RA increases with age until the mid 70s. A prevalence of 0.5-1% is reported in diverse populations world-wide.

Treatments for RA focus on relieving pain, reducing inflammation, slowing or stopping joint damage, and improving patients' well being and ability to function. Current therapies include non-steroidal anti-inflammatory drugs (NSAIDs) which target the clinical features of the disease to alleviate the pain and swelling that accompany RA, disease-modifying anti-rheumatic drugs (DMARDs) which target the actual cause of the disease and biological agents which are genetically engineered to target and modify the autoimmune response. Non-steroidal anti-inflammatory drugs are effective in managing the symptoms of RA, but are limiting as they cannot suppress progression of the disease. First line treatment on confirmation of RA is the use of DMARDs, supported by pain relief medication.

Biologic agents (TNF antagonists, anti B-cell agents and anti-interleukins) have proven effective in RA symptoms management. TNF antagonists have become an important therapeutic option in the treatment of advanced RA.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with RA based on the ARA 1987 revised criteria at least 16 weeks prior to study enrolment, Day 0
* Have an ACR global functional status class of 1 to 3
* Have active disease, defined as the presence of 6 swollen joints and 6 tender joints in a 44 joint examination
* Have a CRP level at screening of ≥ 1.5 mg/dL
* Have been taking oral or parenteral methotrexate (15 mg weekly or above), have been using methotrexate for at least 16 weeks (up to Day 0 of study), and have been on a stable dose for at least 8 weeks, up to Day 0.

Exclusion Criteria:

* Arthritis onset prior to 16 years old
* Any of the following infections:
* Known or acute infection that may affect CRP levels
* Active tuberculosis
* Known chronic infection with human immunodeficiency virus (HIV), hepatitis C virus (HCV) or hepatitis B virus (HBV) including positive serology
* Ongoing systemic inflammatory condition which may interfere with the results of clinical or laboratory tests planned in the study (eg, systemic lupus erythematosus or any other systemic rheumatic disease other than RA)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2007-10; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy (ACR20) of Rob 803 administered orally once daily for 12 weeks in combination with a stable dose of methotrexate in subjects with moderate or severe active RA. | 12 weeks

SECONDARY OUTCOMES:
Evaluate the safety of Rob 803 administered orally once daily in combination with a stable dose of methotrexate in subjects with moderate or severe active RA | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lars Klareskog, Professor, Principal Investigator — Karolinska University Hospital
Locations (34):
- Belgium (3):
  - CUB Hôpital Erasme Université Libre de Bruxelles Service de Rhumatologie, Brussels
  - AZ Sint-Lucas Gent Reumatologie, Ghent
  - Reumainstituut Anne Frankplein 17, Hasselt
- Bulgaria (5):
  - Clinic of Cardiology and Rheumatology UMHAT "Dr. Georgi Stranski", Pleven
  - UMHAT sveti georgi, Ploviv
  - Clinic of Rheumatology MHAT "Sveti Ivan Rilski", Sofia
  - Department of Rheumocardiology, Pulmonology and General Therapy, Sofia
  - Clinic of Rheumatology, UMHAT "Sveta Marina",, Varna
- Georgia (2):
  - Academician V Tsitlanadze Scientific-Practical Centre of Rheumatolgoy, Tbilisi
  - Rheumatology Department Cemotherapy and Immunotherapy Clinical, Tbilisi
- Latvia (2):
  - D Saulites-Kandevicas gimenes arsta prakse, Liepāja, Aldaru Iela 8,
  - Salenieces arsta reimatologa prakse, Valmiera
- Lithuania (3):
  - Rheumatology Clinic Hospital of Kaunas University of Medicine, Kaunas
  - Department of Therapy and diagnostics Siauliai district hospital, Šiauliai
  - Center of Reumathology Vilnius University hospital Santariskiu Clinics, Vilnius
- Poland (6):
  - Centrum Miriada Prywatny Gabinet, Bialystok
  - Szpital Specjalistyczny Nr 1 Oddzial Reumatologii i Rehabilitacji, Bytom
  - Poznanski Osrodek Medyczny Nova Med, Poznan
  - Indywidualna Specjalistyczna Praktyka, Szczecin
  - Centrum Medyczne Osteomed, Warsaw
  - Prywatny Gabinet Lekarski, Wroclaw
- Romania (6):
  - "Sf. Maria" Clinical Hospital, Bucharest
  - "Dr. I. Cantacuzino" Clinical Hospital, Bucharest
  - Emergency Clinical County Hospital, Cluj-Napoca
  - "Dr. Constantin Papilian", Cluj-Napoca
  - Rehabilitation Clinical Hospital, Lasi
  - Emergency County Hospital, Sibiu
- Serbia (2):
  - Institute of Rheumatology Belgrade, Belgrade
  - Institute for Prevention, Treatment and Rehabilitation of Rheumatic and Cardiovascular Diseases, Niška Banja
- Reumatologiska kliniken Karolinska Sjukhuset, Stockholm, Sweden
- United Kingdom (4):
  - Musculo Skeletal dept Chapel Allerton Hospital, Leeds
  - Vectasearch Clinic Ltd St Mary's Hospital, Newport
  - Rheumatology Unit North Tyneside District General Hospital, North Shields
  - Norfolk and Norwich University Hospital, Norwich